CLINICAL TRIAL: NCT06384352
Title: A Phase 1, Multicenter, Open-Label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of YL211 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study to Evaluate the Safety,Tolerability, Pharmacokinetics, and Efficacy of YL211 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL211-INT-101-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-25 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose-Escalation Part (Experimental): Dose-Escalation Part
  Interventions: Drug: YL211
- Part 2: Backfill Enrollment Part (Experimental): Backfill Enrollment Part
  Interventions: Drug: YL211
- Part 3: Dose-Expansion Part (Experimental): Dose-Expansion Part
  Interventions: Drug: YL211

INTERVENTIONS:
Drug: YL211 — Patients will be treated with YL211 intravenous (IV) infusion.

SUMMARY:
This is a multicenter, open-label, Phase 1 study. The study will enroll subjects with advanced solid tumors. It consists of three parts. Part 1 is dose-escalation part. In part 1, the safety and tolerability of YL211 in patients with selected advanced solid tumors will be evaluated and the MTD and RED will be determined.

Part 2 is backfill enrollment part. We will further estimate the safety and efficacy of YL211 in patients with selected adcance tumor to select the RED(s) of YL211.

Part 3 is dose-expansion part. In this part, we will further evaluate the safety and efficacy of YL211 at the MTD/RED(s) in patients with selected advanced solid tumors YL211 will be administered intravenously (IV) until criteria of treatment discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the trial before the start of the trial and voluntarily sign their name and date on the ICF.
2. Aged ≥18 years.
3. Be able and willing to comply with protocol visits and procedures.
4. History of an advanced solid tumors who failed currently available standard therapies and are not amenable to surgical resection, or for whom no available standard therapy or no other approved therapeutic options that have demonstrated clinical benefit.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
6. Adequate organ and bone marrow function.
7. Have at least 1 extracranial measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Exclusion Criteria:

1. Inadequate washout period for prior anticancer treatment before the first dose of study drug.
2. Uncontrolled or clinically significant cardiovascular and cerebrovascular diseases.
3. Clinically significant concomitant pulmonary disease.
4. Uncontrolled infection that requires systemic therapy within 2 weeks before the first dose.
5. Unresolved toxicities from previous anticancer therapy.
6. A history of severe hypersensitivity reactions to the drug substances, inactive ingredients in the drug product, or other monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2029-04-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate nature and frequency of AEs of YL211 in patients with advanced solid tumors according to NCI CTCAE version 5.0 | Approximately within 36 months
  adverse events (AEs)
To evaluate nature and frequency of DLTs in part 1. | Approximately within 36 months
  dose-limiting toxicity (DLT)
ORR assessed using RECIST version 1.1 | Approximately within 36 months
  Objective Response Rate
To determine the MTD and select the recommended expansion dose(s) (RED(s)) of YL211 in patients with advanced solid tumors | Approximately within 36 months
  maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
To characterize the AUC of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  area under the curve (AUC)
To characterize the Cmax of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  maximum concentration (Cmax)
To characterize the Ctrough of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  trough concentration (Ctrough)
To characterize the Tmax of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  time of maximum observed concentration (Tmax)
To characterize the CL of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  clearance (CL)
To characterize the Vd of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  volume of distribution (Vd)
To characterize the t1/2 of YL211 antibody-drug conjugate, YL211 total antibody, unconjugated payload | Approximately within 36 months
  half-life time (t1/2)
To evaluate the anti-drug immune response after treatment with YL211 | Approximately within 36 months
To evaluate DCR of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  disease control rate(DCR, the sum of CR rate, PR rate, and stable disease [SD] rate)
To evaluate DoR of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  duration of response (DoR)
To evaluate SD of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  stable disease(SD)
To evaluate TTR of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  time to response (TTR)
To evaluate PFS of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  progression free survival (PFS)
To evaluate OS of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months
  overall survival (OS)
To evaluate percent change in target lesion of YL211 in patients with advanced solid tumors using RECIST version 1.1 | Approximately within 36 months

OTHER OUTCOMES:
Characterization of genomic alterations that are predictive of response to YL211 | Approximately within 36 months
The use of circulating tumor DNA (ctDNA) to monitor response to YL211 treatment | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (11):
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Sarah Cannon Research Institute (SCRI) at HealthONE, Denver, Colorado
  - Yale School of Medicine - Yale Cancer Center - Smilow Cancer Hospital Care Centers - North Haven, North Haven, Connecticut
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - Sarasota Cattlemen Office, Sarasota, Florida
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - University of Cincinnati Vontz Center for Molecular Studies, Cincinnati, Ohio
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology - Houston, Houston, Texas
  - NEXT Oncology - Dallas, Irving, Texas
  - NEXT San Antonio, San Antonio, Texas
- Australia (3):
  - Gosford Hospital, Gosford, New South Wales
  - One Clinical Research - Nedlands, Nedlands, Western Australia
  - Monash Health, Melbourne
- Canada (2):
  - Princess Margaret Hospital, Toronto, Toronto
  - The Ottawa Hospital - General Campus, Ottawa
- China (5):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Wenzhou Medical University - The First Affiliated Hospital, Wenzhou, Zhejiang
  - West China Hospital, Sichuan University, Chengdu
  - Sun Yat-sen University Cancer Center, Guangzhou